CLINICAL TRIAL: NCT06959602
Title: Antibacterial Efficacy and Outcomes of Root Canal Irrigation Methods
Acronym: ENDOABG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Giorgos Tzanetakis, Associate Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 691/18.02.2025; Giorge Tzanetakis (Other: National and Kapodistrian University of Athens)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Pulp Necrosis; Apical Periodontitis; Endodontic Treatment
Keywords: Quantitative PCR (qPCR); Intracanal Bacteria; XP-Endo Finisher; Passive Ultrasonic Irrigation (PUI); Sodium Hypochlorite
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The operator performing the procedure is not blinded, but outcome assessors evaluating healing at follow-up could be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Final Irrigation with 2.5% Sodium Hypochlorite (Other): Root canals will be irrigated with 2.5% sodium hypochlorite as the final irrigation without activation.
  Interventions: Procedure: Final Irrigation with 2.5% Sodium Hypochlorite
- Passive Ultrasonic Irrigation with NaOCl (Other): Root canals will be irrigated with 2.5% sodium hypochlorite activated by Passive Ultrasonic Irrigation (PUI).
  Interventions: Procedure: Passive Ultrasonic Irrigation (PUI) with Sodium Hypochlorite
- XP-Endo Finisher activation with NaOCl (Other): Root canals will be irrigated with 2.5% sodium hypochlorite followed by mechanical activation using the XP-Endo Finisher file.
  Interventions: Procedure: XP-Endo Finisher Activation with Sodium Hypochlorite

INTERVENTIONS:
Procedure: Final Irrigation with 2.5% Sodium Hypochlorite — After supragingival scaling and removal of caries or defective restorations, the tooth will be isolated and disinfected with 3% H202 and 2.5% NaOCl. Access preparation will be done using a sterile high-speed bur under sterile saline irrigation, followed by re-disinfection. NaOCl will be neutralized with 5% sodium thiosulphate, and sterility will be confirmed via paper point sampling. Only teeth with negative sterility samples will proceed. Sample S1 will be collected after saline irrigation and mild instrumentation with a sterile K-file #15, using an apex locator. Paper points will absorb canal fluid and be frozen in Tris-EDTA buffer at -20°C. Complete chemomechanical preparation will follow, with irrigation after each instrument change. Cervical and mid-thirds will be enlarged with Gates-Glidden burs and the apical third with NiTi RaCe files (40/04). Sample S2 will be taken after preparation. Group A will receive final irrigation with 2.5% NaOCl before collection of sample S3.
  Other Names: NaOCl 2.5%
  Arms: Final Irrigation with 2.5% Sodium Hypochlorite
Procedure: Passive Ultrasonic Irrigation (PUI) with Sodium Hypochlorite — Activation of 2.5% sodium hypochlorite solution inside the root canal system using Passive Ultrasonic Irrigation (PUI) after chemomechanical preparation. Group B, sample (S3).
  Other Names: PUI; Ultrasonic Activation; Passive Ultrasonic Irrigation
  Arms: Passive Ultrasonic Irrigation with NaOCl
Procedure: XP-Endo Finisher Activation with Sodium Hypochlorite — Mechanical activation of 2.5% sodium hypochlorite solution using the XP-Endo Finisher instrument following chemomechanical preparation.Group C, sample (S3).
  Other Names: XP-Endo Finisher; XPF Activation
  Arms: XP-Endo Finisher activation with NaOCl

SUMMARY:
This randomized clinical trial aims to evaluate the antibacterial efficacy and treatment outcomes of three different final irrigation protocols during root canal therapy: 2.5% sodium hypochlorite alone, sodium hypochlorite with Passive Ultrasonic Irrigation (PUI), and sodium hypochlorite with XP-Endo Finisher activation. Sixty-six single-rooted teeth with pulp necrosis and apical periodontitis will be randomly assigned to one of the three groups. Antibacterial efficacy will be assessed through Real-Time PCR quantification of total bacterial load and four specific bacterial species before and after treatment. Treatment success will be evaluated clinically and radiographically at 6 and 12 months. The study aims to identify the most effective irrigation strategy for bacterial reduction and healing outcomes.

DETAILED DESCRIPTION:
This randomized, two-arm, parallel clinical trial investigates the antibacterial effectiveness and clinical outcomes of three root canal final irrigation protocols in teeth with pulp necrosis and apical periodontitis. Following standard chemomechanical preparation, participants' teeth will be randomly assigned to one of three interventions: final irrigation with 2.5% sodium hypochlorite alone, sodium hypochlorite activated by Passive Ultrasonic Irrigation (PUI) or sodium hypochlorite activated with the XP-Endo Finisher file.

The study focuses on the reduction of total bacterial load and specific pathogenic bacterial species (Pseudoramibacter alactolyticus, Treponema denticola, Streptococcus anginosus, and Porphyromonas endodontalis ) assessed through highly sensitive quantitative Real-Time PCR analysis of samples collected at different treatment stages. Sampling procedures ensure strict aseptic conditions and standardized protocols for DNA extraction and analysis.

All participants will undergo a standardized endodontic treatment protocol by a single operator to minimize variability. Follow-up includes clinical and radiographic examinations at 6 and 12 months, with healing assessed through the Periapical Index (PAI) and presence or absence of clinical symptoms.

This trial aims to provide new clinical evidence regarding the added value of supplementary irrigation techniques, comparing their ability to reduce bacterial burden and influence long-term treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the patients who wish to participate in the study.
* Single-rooted teeth with pulp necrosis confirmed by pulp sensibility tests, negative response to both cold and electric pulp testing and radiographic evidence of apical periodontitis.
* Teeth with relatively straight canals, complete root development and no radiographic evidence of pulp canal obliteration.

Exclusion Criteria:

* Patients who have received antibiotic treatment the last 3 months or need chemoprophylaxis for dental treatment.
* Teeth with previous endodontic treatment.
* Teeth with cracks or incomplete vertical root fracture which disturbs the integrity of the pulp chamber walls or teeth with the pulp chamber exposed to oral environment.
* Teeth with periodontal pocket more than 4mm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Total Intracanal Bacterial Load | 0ne to six months
  Quantitative reduction of the total intra canal bacterial load measured by Real-Time PCR (qPCR) after final irrigation procedures.

SECONDARY OUTCOMES:
Reduction in Specific Bacterial Species | one to six months
  Quantitative change of Pseudoramibacter alactolyticus, Treponema denticola, Streptococcus anginosus, and Porpyromonas endodontalis measured by Real-Time PCR after supplementary irrigation procedures.
Clinical and Radiographic Healing Outcome | 6 months and 12 months after root canal treatment
  Healing of periapical lesions assessed clinically and radiographically (using the Periapical Index, PAI) at 6 and 12 months after treatment.

OTHER OUTCOMES:
Comparison of Antibacterial Effectiveness Between Interventions | Immediately post-treatment and at 12 months follow-up
  Comparison of the bacterial load reduction and treatment success rates among the three irrigation strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Giorge Tzanetakis, Dr (PhD), Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
The IPD that will be shared include anonymized data related to the bacterial load measurements (qPCR results for total bacterial load and for Pseudoramibacter alactolyticus, Treponema denticola, Streptococcus anginosus, and Porphyromonas endodontalis), treatment group allocation (NaOCl 2.5% only, NaOCl 2.5% + Passive Ultrasonic Irrigation (PUI), or NaOCl 2.5% + XP Endo Finisher), and treatment outcomes based on clinical and radiographic follow-up (e.g., PAI scores, presence/absence of clinical signs and symptoms).
  No data containing directly identifiable patient information (e.g., names, personal identification numbers) will be shared.
  The data will be available upon reasonable request to the principal investigator after the publication of the study results, with the requirement of a data-sharing agreement to ensure appropriate use. The sharing will comply with ethical approvals and participants' consent agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The individual participant data (IPD) and supporting documents will become available starting 6 months after the publication of the main study results. Data will be available for a minimum of 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound research proposal and agree to a data-sharing agreement will be eligible to access the data. Proposals will be reviewed by the study's advisory committee to ensure they are appropriate and ethical. Access will be granted for academic, non-commercial research purposes only. Data will be provided through a secure platform ensuring confidentiality and data protection.

REFERENCES:
- [Result] Orstavik D. Root canal disinfection: a review of concepts and recent developments. Aust Endod J. 2003 Aug;29(2):70-4. doi: 10.1111/j.1747-4477.2003.tb00515.x. PMID 14655819
- [Result] Siqueira JF Jr, Rocas IN. Clinical implications and microbiology of bacterial persistence after treatment procedures. J Endod. 2008 Nov;34(11):1291-1301.e3. doi: 10.1016/j.joen.2008.07.028. Epub 2008 Sep 17. PMID 18928835
- [Result] Luciano Giardino, Marco Morra, Carlo Becce, Fernanda G. Pappen, Zahed Mohammadi, Flavio Palazzi,Comparative wettability of different sodium hypochlorite solutions,Giornale Italiano di Endodonzia.2012; 26(22):1121-4171 doi:org/10.1016/j.gien.2012.06.002.
- [Result] Weber CD, McClanahan SB, Miller GA, Diener-West M, Johnson JD. The effect of passive ultrasonic activation of 2% chlorhexidine or 5.25% sodium hypochlorite irrigant on residual antimicrobial activity in root canals. J Endod. 2003 Sep;29(9):562-4. doi: 10.1097/00004770-200309000-00005. PMID 14503827
- [Result] Mohammadi Z, Abbott PV. Antimicrobial substantivity of root canal irrigants and medicaments: a review. Aust Endod J. 2009 Dec;35(3):131-9. doi: 10.1111/j.1747-4477.2009.00164.x. PMID 19961451
- [Result] Ricucci D, Siqueira JF Jr, Bate AL, Pitt Ford TR. Histologic investigation of root canal-treated teeth with apical periodontitis: a retrospective study from twenty-four patients. J Endod. 2009 Apr;35(4):493-502. doi: 10.1016/j.joen.2008.12.014. PMID 19345793
- [Result] Sjogren U, Figdor D, Persson S, Sundqvist G. Influence of infection at the time of root filling on the outcome of endodontic treatment of teeth with apical periodontitis. Int Endod J. 1997 Sep;30(5):297-306. doi: 10.1046/j.1365-2591.1997.00092.x. PMID 9477818
- [Result] Sjogren U, Hagglund B, Sundqvist G, Wing K. Factors affecting the long-term results of endodontic treatment. J Endod. 1990 Oct;16(10):498-504. doi: 10.1016/S0099-2399(07)80180-4. PMID 2084204
- [Result] Paixao S, Rodrigues C, Grenho L, Fernandes MH. Efficacy of sonic and ultrasonic activation during endodontic treatment: a Meta-analysis of in vitro studies. Acta Odontol Scand. 2022 Nov;80(8):588-595. doi: 10.1080/00016357.2022.2061591. Epub 2022 Apr 17. PMID 35430959
- [Result] Mancini M, Cerroni L, Iorio L, Armellin E, Conte G, Cianconi L. Smear layer removal and canal cleanliness using different irrigation systems (EndoActivator, EndoVac, and passive ultrasonic irrigation): field emission scanning electron microscopic evaluation in an in vitro study. J Endod. 2013 Nov;39(11):1456-60. doi: 10.1016/j.joen.2013.07.028. Epub 2013 Sep 6. PMID 24139274
- [Result] Alves FR, Marceliano-Alves MF, Sousa JC, Silveira SB, Provenzano JC, Siqueira JF Jr. Removal of Root Canal Fillings in Curved Canals Using Either Reciprocating Single- or Rotary Multi-instrument Systems and a Supplementary Step with the XP-Endo Finisher. J Endod. 2016 Jul;42(7):1114-9. doi: 10.1016/j.joen.2016.04.007. Epub 2016 May 20. PMID 27215810
- [Result] Matoso FB, Quintana RM, Jardine AP, Delai D, Fontanella VRC, Grazziotin-Soares R, Kopper PMP. XP Endo Finisher-R and PUI as supplementary methods to remove root filling materials from curved canals. Braz Oral Res. 2022 Apr 15;36:e053. doi: 10.1590/1807-3107bor-2022.vol36.0053. eCollection 2022. PMID 35442382
- [Result] Poly A, Marques F, Lee J, Setzer FC, Karabucak B. XP-endo Finisher effectively reduces hard-tissue debris accumulated in root canals with isthmus after preparation with a reciprocating file system. Aust Endod J. 2023 Aug;49(2):279-286. doi: 10.1111/aej.12676. Epub 2022 Aug 18. PMID 35980742
- [Result] de Jesus Oliveira LS, de Figueiredo FED, Dantas JA, Ribeiro MAG, Estrela C, Sousa-Neto MD, Faria-E-Silva AL. Impact XP-endo finisher on the 1-year follow-up success of posterior root canal treatments: a randomized clinical trial. Clin Oral Investig. 2023 Dec;27(12):7595-7603. doi: 10.1007/s00784-023-05349-9. Epub 2023 Oct 23. PMID 37867163
- [Result] Amaral RR, Guimaraes Oliveira AG, Braga T, Reher P, de Macedo Farias L, Magalhaes PP, Ferreira PG, Ilma de Souza Cortes M. Quantitative Assessment of the Efficacy of Two Different Single-file Systems in Reducing the Bacterial load in Oval-Shaped Canals: A Clinical Study. J Endod. 2020 Sep;46(9):1228-1234. doi: 10.1016/j.joen.2020.06.007. Epub 2020 Jul 9. PMID 32653532
- [Result] Ballal NV, Gandhi P, Shenoy PA, Dummer PMH. Evaluation of various irrigation activation systems to eliminate bacteria from the root canal system: A randomized controlled single blinded trial. J Dent. 2020 Aug;99:103412. doi: 10.1016/j.jdent.2020.103412. Epub 2020 Jun 22. PMID 32585261
- [Result] Tzanetakis GN, Koletsi D, Tsakris A, Vrioni G. Prevalence of Fungi in Primary Endodontic Infections of a Greek-living Population Through Real-time Polymerase Chain Reaction and Matrix-assisted Laser Desorption/Ionization Time-of-flight Mass Spectrometry. J Endod. 2022 Feb;48(2):200-207. doi: 10.1016/j.joen.2021.11.003. Epub 2021 Nov 17. PMID 34800484
- [Result] Coaguila-Llerena H, Ordinola-Zapata R, Staley C, Dietz M, Chen R, Faria G. Multispecies biofilm removal by a multisonic irrigation system in mandibular molars. Int Endod J. 2022 Nov;55(11):1252-1261. doi: 10.1111/iej.13813. Epub 2022 Aug 30. PMID 35976101
- [Result] Lima AR, Herrera DR, Francisco PA, Pereira AC, Lemos J, Abranches J, Gomes BPFA. Detection of Streptococcus mutans in symptomatic and asymptomatic infected root canals. Clin Oral Investig. 2021 Jun;25(6):3535-3542. doi: 10.1007/s00784-020-03676-9. Epub 2020 Nov 10. PMID 33170373
- [Result] Siqueira JF Jr, Rocas IN. Pseudoramibacter alactolyticus in primary endodontic infections. J Endod. 2003 Nov;29(11):735-8. doi: 10.1097/00004770-200311000-00012. PMID 14651280
- [Result] Rosa TP, Signoretti FG, Montagner F, Gomes BP, Jacinto RC. Prevalence of Treponema spp. in endodontic retreatment-resistant periapical lesions. Braz Oral Res. 2015;29:S1806-83242015000100228. doi: 10.1590/1807-3107BOR-2015.vol29.0031. Epub 2015 Jan 27. PMID 25627883
- [Result] Ordinola-Zapata R, Costalonga M, Dietz M, Lima BP, Staley C. The root canal microbiome diversity and function. A whole-metagenome shotgun analysis. Int Endod J. 2024 Jul;57(7):872-884. doi: 10.1111/iej.13911. Epub 2023 Mar 29. PMID 36861850
- [Result] Ordinola-Zapata R, Costalonga M, Nixdorf D, Dietz M, Schuweiler D, Lima BP, Staley C. Taxonomic abundance in primary and secondary root canal infections. Int Endod J. 2023 Feb;56(2):278-288. doi: 10.1111/iej.13864. Epub 2022 Nov 22. PMID 36334085
- [Result] Rocas IN, Siqueira JF Jr. Comparison of the in vivo antimicrobial effectiveness of sodium hypochlorite and chlorhexidine used as root canal irrigants: a molecular microbiology study. J Endod. 2011 Feb;37(2):143-50. doi: 10.1016/j.joen.2010.11.006. PMID 21238793
- [Result] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Result] Orstavik D. Reliability of the periapical index scoring system. Scand J Dent Res. 1988 Apr;96(2):108-11. PMID 3162597
- [Result] Kirkevang LL, Orstavik D, Wenzel A, Vaeth M. Prognostic value of the full-scale Periapical Index. Int Endod J. 2015 Nov;48(11):1051-8. doi: 10.1111/iej.12402. Epub 2014 Nov 24. PMID 25354086
- [Result] Kirkevang LL, Orstavik D, Bahrami G, Wenzel A, Vaeth M. Prediction of periapical status and tooth extraction. Int Endod J. 2017 Jan;50(1):5-14. doi: 10.1111/iej.12581. Epub 2015 Dec 23. PMID 26580306

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT06959602/Prot_SAP_003.pdf
  • Informed Consent Form (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT06959602/ICF_004.pdf